CLINICAL TRIAL: NCT03627143
Title: Decreasing Hospital Admissions From the Emergency Department for Acute Atrial Fibrillation
Brief Title: Decreasing Hospital Admissions From the ED for AAFF
Acronym: RAFF-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20180367-01T
Record Dates: First submitted 2018-07-19; First posted 2018-08-13 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Intervention Model Description: Multicentre Behaviour Intervention Trial using a Stepped Wedge Cluster Randomized Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local implementation of AAFF guidelines (Other): The study intervention will support local implementation of the CAEP AAFF Guidelines during the intervention periods of the trial. The investigators will identify behaviour change techniques and organization/system level strategies that could likely address identified barriers or enhance enablers.
  Interventions: Other: KTI activities

INTERVENTIONS:
Other: KTI activities — The Investigators also plan the following activities to encourage adherence to the guidelines, with an ultimate goal of rhythm or rate control and discharge home for most patients.
  1. Selection of one or more local physician champions from both the ED as well as the cardiology group;
  2. Review and discussion of the goals of the study, as well as perceived barriers and enablers, by the ED and cardiology physician groups;
  3. Formal introduction of the CAEP AAFF Guidelines to the ED physicians and residents by means of presentations at rounds and staff meetings, emails, online video, and web-based resources;
  4. Development of local action plan addressing local barriers to implementation;
  5. Provision of the free Smartphone App to be developed for the guidelines;
  6. Regular reminders provided by the local research staff;
  7. Audit and feedback charts of site compliance

SUMMARY:
Acute atrial fibrillation and flutter (AAFF) is characterized by rapid heart rates with onset less than seven days. It's the most common type of palpitation treated in the Emergency Department (ED). Some Canadian ED's will discharge 95% of AAFF patients whereas others admit up to 40%. With hospital and ED crowding, discharge is the most optimal, effective and safe strategy. Our aim is to improve the care and reduce the length of stay (LOS) of ED AAFF patients, while decreasing unnecessary hospitalizations. First, the investigators must understand the local barriers. In the previous study, the investigators conducted interviews of emergency physicians, cardiologists and AAFF patients. In Project 1b, the investigators created the CAEP ED AAFF Guidelines Checklist to assist physicians to manage AAFF more efficiently and safely. The Guidelines are comprised of two algorithms and four sets of checklists for ED assessment and management. They have been endorsed by CAEP and are published in CJEM.

The investigators are now planning Project 2 in which the investigators will conduct a cluster [group] randomized trial at 11 Canadian EDs and enroll 1,300 patients over thirteen months. The investigators are not randomizing individual patients or doctors; instead the investigators are randomizing the start date of individual hospitals. Our goal is to introduce the new Guidelines into these hospitals to improve the care of AAFF patients. The investigators hope to improve AAFF management, leading to a significant decrease in hospital admissions and ED LOS. Central to our plans will be engagement of our two patient partners. Our behaviorally optimized intervention will be developed using state-of-the-art implementation science approaches informed by the results of Project 1a. The investigators will also undertake within-project and end-of-project knowledge translation and implementation (KTI) strategies to facilitate scale up and roll out of our program to ED departments in small, medium, and large hospitals across Canada (future Project 3). Ultimately the investigators expect to improve ED practices and decrease AAFF admissions and LOS, without increasing visits.

ELIGIBILITY:
All eligible patients seen in the participating EDs during the study period will be included in the trial regardless of how they are managed.

Inclusion Criteria:

* stable patients presenting with an episode of acute atrial fibrillation or flutter (AAFF) of at least 3 hours duration, where symptoms require ED management by rhythm or rate control.
* patients with a history of prior episodes of AAFF, or those with previous presentations during the study periods.

Exclusion Criteria: We will exclude patients who have any of the reasons listed below.

* have permanent (chronic) AF
* are deemed unstable and require immediate cardioversion: i) systolic blood pressure <90 mmHg; ii) rapid ventricular pre-excitation (Wolff-Parkinson-White syndrome); iii) acute coronary syndrome - ongoing severe chest pain and marked ST depression (>2mm) on ECG despite therapy; or iv) pulmonary edema - severe dyspnea requiring immediate IV diuretic, nitrates, or BIPAP;
* the primary presentation was for another condition rather than arrhythmia
* convert spontaneously to sinus rhythm prior to receiving physician-initiated therapy; or
* die while in the ED from non-AAFF related causes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
length of stay in ED in minutes | a 100 minute reduction in ED length of stay (or a relative reduction of approximately 25%)
  Length of stay in ED in min. from time of arrival to time of discharge or admission.

SECONDARY OUTCOMES:
Use of rhythm control in the ED | 13 months
  attempts at chemical or electrical cardioversion, as well as the success of these attempts (we believe these attempts facilitate ED discharge); compliance with the AAFF Guidelines will be assessed on criteria to be determined a priori by the investigators;
Use of rate control and the final heart rate at disposition | 13 months
  compliance with the AAFF Guidelines will be assessed on criteria to be determined a priori by the investigators;
Appropriate prescription of anticoagulants on discharge | 1 day
  anticoagulation prescription in compliance with the AAFF Guidelines
Adverse events | 30 days from discharge from the ED
  measuring adverse events within 30 days of discharge from the emergency department
Return ED visits and admission | 30 days
  for AAFF or related cardiovascular problems (stroke, CHF, AAFF, ACS or death), in the subsequent 30 days via a Health record reivew

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stiell, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (12):
- Canada (12):
  - Dr. Georges-L. - Dumont University Hospital, Moncton, New Brunswick
  - Dartmouth General Hospital, Dartmouth, Nova Scotia
  - Ottawa Hospital, Ottawa, Ontario
  - St. Joseph's Health Center, Toronto, Ontario
  - Hopital Du Sacre-Coeur, Montreal, Quebec
  - Hôpital Charles-Lemoyne, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Hôtel-Dieu de Lévis, Québec, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No